CLINICAL TRIAL: NCT05645731
Title: Lung Cancer Screening in Family Members and Peers of Lung Cancer Patients: a Prospective Cohort Study
Status: Completed | Type: Observational
Sponsor: Nicole Ezer, MD, FRCPC, MPH (Other)
Responsible Party: Sponsor-Investigator, Nicole Ezer, MD, FRCPC, MPH, Assistant professor of medicine, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Other Study IDs: MP-37-2023-9041
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Lung Cancer; Lung Cancer Screening; Patient Empowerment
MeSH Terms: conditions — Lung Neoplasms; Patient Participation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Lung cancer patient: Lung cancer patients or lung cancer survivors willing to refer close contacts for lung cancer screening
- Referred participants: Participants referred to the study by close contacts living with lung cancer.

SUMMARY:
Lung cancer screening of active or former heavy smokers with yearly low-dose CT allows for earlier diagnosis and better lung cancer survival. Risk of developing lung cancer is higher among family members and close contacts of lung cancer patients, because of shared genetics, environment and life habits like smoking. The investigators want to engage lung cancer patients to refer their family members and close contacts for lung cancer screening, and evaluate if this referred population have higher risk of lung cancer than the population referred by their family doctors.

ELIGIBILITY:
Lung cancer patients:

Inclusion Criteria:

* > 18 years old
* Current or former lung cancer patient

Exclusion Criteria: none

Referred participants Inclusion criteria: >18 years old Exclusion criteria: Personal history of lung cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Lung cancer patient recruited at clinics at the MUHC.
  2. Close contacts of lung cancer patients referred to our study
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-05-12 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Mean number of referrals for lung cancer screening per participants | 2 weeks post inclusion
  Mean number of referrals for lung cancer screening per participants: lung cancer participants will refer contacts directly on the REDCap questionnaire at enrollment. They will be contacted a second time 2 weeks after enrollment and asked if they referred additional people in their entourage for lung cancer screening.
Mean PLCOm2012 risk prediction model score among referred participants | baseline
  Mean risk of developing lung cancer in the next 6 years using the validated PLCOm2012 risk prediction model in smokers or ex-smokers referred participants that are 55 to 74 years old.

SECONDARY OUTCOMES:
Number of visitors on our website for referred participants | 6 months
  Quantification of people who visited the website for close contacts of lung cancer patients: Number of unique access to website based on google analytics data.
Number of people who started to fill the enrollment form for referred participants. | 6 months
  Number of people who started to fill the enrollment form for referred participants.
Number of referred participants who enrolled in the study. | 6 months
  Number of referred participants who enrolled in the study.
PLCO score as a binary outcome (above or below 2%) among referred participants | baseline
Proportion of LCS eligible participants who will complete lung cancer screening within 18 months of referral by a lung cancer patient | 18 months
  Proportion of LCS eligible participants who will complete lung cancer screening within 18 months of referral by a lung cancer patient
Proportion of individuals who would theoretically demonstrate interest in genetic testing to assess for lung cancer risk. | baseline
  Proportion of individuals who would theoretically demonstrate interest in genetic testing to assess for lung cancer risk.
Proportion of individuals who demonstrate interest in referral to a smoking cessation program among referred participants that are current smokers | baseline
  Proportion of individuals who demonstrate interest in referral to a smoking cessation program among referred participants that are current smokers
Anxiety regarding lung cancer for referred participants | baseline
  GAD7
Anxiety regarding lung cancer for referred participants | 1 month
  GAD7

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Ezer, MD, Principal Investigator — Research Institute of the McGill University Health Center
Locations (1):
- MUHC, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Pitrou I, Petrangelo A, Besson C, Pepe C, Waschke AH, Agulnik J, Gonzalez AV, Ezer N. Lung Cancer Screening in Family Members and Peers of Patients With Lung Cancer: Protocol for a Prospective Cohort Study. JMIR Res Protoc. 2025 Mar 28;14:e58529. doi: 10.2196/58529. PMID 40153794